CLINICAL TRIAL: NCT02479048
Title: The Impact of Avocado Fruit on Postprandial Markers of the Glycemic Response, Satiety/Appetite and Cardiometabolic Risk: An Acute Dose Response Study
Brief Title: Avocado Fruit on Postprandial Markers of the Glycemic Response, Satiety/Appetite and Cardiometabolic Risk
Acronym: AVOC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB2015-001
Record Dates: First submitted 2015-06-19; First posted 2015-06-23 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Glycemic Response
Keywords: satiety/appetite; glycemic response; cardiometabolic risk

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test meal 1 (TM1) (Active Comparator): High fat meal (HF) with ½ avocado (~68g)
  Interventions: Dietary Supplement: Test meal 1
- Test meal 2 (TM2) (Active Comparator): High fat meal (HF) with 1 avocado (~136g)
  Interventions: Dietary Supplement: Test meal 2
- Control meal (CM) (Placebo Comparator): High carbohydrate, high saturated fat control meal (CM) without avocado.
  Interventions: Dietary Supplement: Control Meal (CM)

INTERVENTIONS:
Dietary Supplement: Test meal 1 — High fat meal (HF) with ½ avocado (~68g), matched to CM for energy content; not matched for macronutrient content or type (e.g., fat type).
  Arms: Test meal 1 (TM1)
Dietary Supplement: Test meal 2 — High fat meal (HF) with 1 avocado (~136g) matched for energy but not macronutrient content or type.
  Arms: Test meal 2 (TM2)
Dietary Supplement: Control Meal (CM) — High carbohydrate, high saturated fat control meal (CM) without avocado.
  Arms: Control meal (CM)

SUMMARY:
The primary goal is to characterize the acute effects of avocado intake on glycemic and satiety/ appetite responses in relatively healthy overweight / obese adults. The secondary goal is to investigate risk factors for cardio-metabolic disease.

DETAILED DESCRIPTION:
The trial is a single center randomized, 3-arm, controlled, within-subject crossover study utilizing a multiple sampling, repeated measures paradigm. The trial will test 3 treatment conditions in 30 relatively healthy men and women 25-60 years of age. Study treatments include Control (without avocado), Test Meal 1 (1/2 avocado; ~68g), and Test Meal 2 (1 Avocado; ~136g).

Subjects will be required to meet several inclusion and exclusion criteria, which will be assessed through online and clinic mechanisms, including questionnaires, blood analysis and anthropometric measures. Eligible subjects will be invited to participate in the study. Each subject will be asked to come for one Information Session/Screening Visit, one Pre-Study Visit, three dinner pick-ups (the day before each test day visit) and three Test Day Visits. Subjects will be randomized to receive test treatments based on randomization schedule at the Pre-Study Visit.

During the Pre-Study Visit subjects will be instructed on the process for completing study questionnaires and counseled to restrict avocado intake and intake of colored plant foods rich in phytonutrients the 3 days prior to each Test Day Visit. They will be asked to restrict alcohol intake, coffee/tea/ caffeinated beverage intake and moderate / vigorous physical activity and to drink plenty of water to maintain hydration in the 24 h prior to each Test Day Visit. They will be instructed to come to the CNRC the day before each Test Day Visit to pick up their dinner meal and evening snack. Subjects will be asked to get at least 7 hours sleep and to come to the CNRC after an overnight fast of 10 h on each Test Day Visit.

Each Test Day Visit will require subjects to be in the clinic for ~7 h to complete all baseline and post challenge meal testing procedures. Subjects will be evaluated for compliance with the protocol (diet, exercise, sleep, fasting), have their body weight and blood pressure measured and baseline flow mediated dilation (FMD) will be recoded before placement of a catheter and baseline blood sample is taken. Baseline subjective satiety will be measured by visual analogue scale (VAS) just before consuming one of the 3 breakfast treatment meals. FMD will be measured at 2 time points after breakfast and blood samples and VAS questionnaires will be collected at multiple time points over the 6 h postprandial period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 25-60 yrs.
* BMI of 25 - 35 kg/m2
* No clinical evidence / history of cardiovascular, respiratory, renal, gastrointestinal, or hepatic disease
* Not taking over-the-counter or prescription medications / dietary supplements that may interfere with study procedures or endpoints (e.g., antioxidant supplements, anti-inflammatory, lipid-lowering or blood pressure lowering medications.
* Fasting blood glucose of 90-115 mg/dl
* Fasting insulin < 13 U/L
* Non-smoker or past smoker (smoking cessation > 2 yrs.)
* has at least 1 large, sturdy and well anchored vein in order to place a catheter

Exclusion Criteria:

* Aged < 25 or > 60 years
* BMI < 25 kg/m2 or > 35 kg/m2
* History of cardiovascular, respiratory, renal, gastrointestinal or hepatic disease
* Diabetes
* Uncontrolled blood pressure (>140 / 90 mmHg)
* Have or had cancer other than non-melanoma skin cancer in past 5 years
* Taking over-the-counter or prescription medications or dietary supplements that may interfere with study procedures or endpoints (including protein powers, energy drinks)
* Fasting blood glucose <90 or > 115 mg/dl
* Fasting insulin ≥ 13 U/L
* Vegan dietary habits, unusual dietary habits or sensitive or allergic to any of the test meal components / ingredients
* Dislike avocados or non-consumers of avocados
* Current smoker
* Actively losing weight or trying to lose weight
* Drug or alcohol addiction
* Present with significant psychiatric or neurological disturbances
* Pregnant, lactating or planning to become pregnant
* Consuming 3 or more servings nuts or peanuts per week
* has no accessible vein site for placing a catheter

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in postprandial blood glucose concentration response for treatments compared to control over 6-hour postprandial period | Baseline to 6 hours
  postprandial blood glucose concentration response

SECONDARY OUTCOMES:
Changes in postprandial endothelial function using Flow Mediated Dilation (FMD) for treatments compared to control | Baseline to 6 hours
  postprandial endothelial function using Flow Mediated Dilation (FMD)
Change in postprandial blood insulin and triglycerides concentration response for treatments compared to control over 6-hour postprandial period | Baseline to 6 hours
  postprandial blood insulin and triglycerides concentration response
Changes in postprandial subjective satiety responses using visual analog scales (VAS) for treatments compared to control over 6-hour postprandial period | Baseline to 6 hours
  postprandial subjective satiety responses using visual analog scales (VAS)
Changes in postprandial gut hormones related to satiety for treatments compared to control over 6-hour postprandial period | Baseline to 6 hours
  postprandial gut hormones related to satiety for treatments

OTHER OUTCOMES:
Changes in postprandial lipoproteins responses for treatments compared to control | Baseline to 6 hours
  postprandial lipoproteins responses
Changes in postprandial inflammation responses for treatments compared to control | Baseline to 6 hours
  postprandial inflammation responses
Changes in postprandial oxidation responses for treatments compared to control | Baseline to 6 hours
  postprandial oxidation responses

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States